CLINICAL TRIAL: NCT05016830
Title: Effect of the Combination of tDCS and Visual Occlusion Therapy on Visual Acuity, Contrast Vision and Depth Vision, in Adult Patients With Amblyopia
Brief Title: Bilateral Transcranial Direct Current Stimulation and Ocular Occlusion for Adults With Amblyopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lock-down in the city of Santiago due to Covid-19 pandemia. Most faculty premises were closed for research purposes and mobility in the city was restricted.
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Romulo Antonio Fuentes Flores, Assistant Professor at Department of Neuroscience, and Director of Research at the Faculty of Medicine of University of Chile, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CECI-HCUCH Nº44-2019
Record Dates: First submitted 2021-08-13; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Amblyopia
Keywords: Lazy eye syndrome; Transcranial direct current stimulation; Ocular occlusion; Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: A randomized, controlled pilot trial, that consists in two groups: a control group that receives sham stimulation and ocular occlusion, and a second group that receives bilateral transcranial direct current stimulation and ocular occlusion.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both sham and bilateral transcranial direct current stimulation were applied with the same electrode configuration, but the functioning of the stimulation device was blinded to the patient, the care provider, and the researcher performing measurements. The operator of the stimulation device selected the stimulation protocol. Sham stimulation protocol consisted of current ramp and delivery of current for 30 seconds and 19 minutes and 30 seconds with no current delivery. Actual stimulation consisted of a current ramp and 20 minutes of current delivery. There were no visual cues allowing to differentiate sham and stimulation protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham bilateral transcranial direct current stimulation (Sham Comparator): Sham bilateral transcranial direct current stimulation consisted of 2 milliamperes (mA) of current from the anodal electrode in the amblyopic primary visual cortex to the cathodal electrode located in the fellow primary visual cortex, but the stimulation was turned off after 30 seconds. On Sham Stimulation onset, the participant's fellow eye was occluded and the participant performed a reading task for 20 minutes.
  Interventions: Device: Bilateral transcranial direct current stimulation
- Bilateral transcranial direct current stimulation (Experimental): Bilateral transcranial direct current stimulation consisted of 2 mA of current from the anodal electrode in the amblyopic primary visual cortex to the cathodal electrode located in the fellow primary visual cortex and the stimulation was on for 20 minutes. On stimulation onset, the participant's fellow eye was occluded and the participant performed a reading task for 20 minutes.
  Interventions: Device: Bilateral transcranial direct current stimulation

INTERVENTIONS:
Device: Bilateral transcranial direct current stimulation — A direct current is applied with two electrodes (cathode and anode) in specific parts of the skull. In this case the anode was over the occipital area to target the amblyopic cortex, while the cathode was over the contralateral side, targeting the fellow cortex.

SUMMARY:
A prospective interventional study is expected to be conducted, to test a possible new treatment for amblyopia (lazy eye syndrome). Bilateral transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation, which may help in visual function recovery of adult patients with amblyopia. This pilot study will test the feasibility of said therapy, along with the short term effects of bilateral tDCS in visual function.

DETAILED DESCRIPTION:
Theoretical Framework: Ocular occlusion treatment has been used classically and with excellent results for the treatment of amblyopia in those under 14 years of age, since in this period it has been seen that there is greater neuroplasticity, leaving little to do in the period of lower neuroplasticity, in young and adult patients with later diagnoses. Transcranial Direct Current Stimulation therapy is an emergent technique used in neurological diseases to increase neuroplasticity, by changing the resting potential of neurons. Our hypothesis is that the combination of tDCS and visual occlusion therapy is capable of increasing visual acuity, contrast sensitivity, and depth perception, in young people over 18 years of age.

Methodology: The application of a double-blind, randomized clinical trial is proposed to evaluate the application of 2 different therapies: Occlusion with bilateral tDCS, and Occlusion with tDCS sham (sham). The study subjects will be randomly assigned to a group, and one session of stimulation will be performed. Data will be analyzed using Student's t test, or Mann-Whitney test, according to the normal or non-normal distribution of the sample, respectively. Also, the change over time of the variables will be measured using the Conditional Change Model.

Expected Results: The investigators expect that visual acuity, contrast vision, and dichoptic vision in the Occlusion therapy group with bilateral tDCS will be significantly higher than the Occlusion therapy group with tDCS sham (sham).

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of Amblyopia

Exclusion Criteria:

* Ophthalmologic disease other than amblyopia
* Chronic pharmacological therapy
* Implanted medical device
* Neurologic disease or surgery history
* History of an adverse reaction to tDCS
* Pregnancy
* Not able to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 1-2 hours
  Clarity or Sharpness in vision, measured in LogMar
Visual Sensitivity | 1-2 hours
  The ability to perceive differences between an object and its background, measured in percentage of contrast sensitivity.
Stereopsis | 1-2 hours
  the perception of depth produced by the reception in the brain of visual stimuli from both eyes in combination. Measured in degrees of arc.
Visual evoked potentials | 1-2 hours
  The electroencephalographic response from the primary visual cortex to a stimuli. Measured in millivolts (mV).

CONTACTS AND LOCATIONS:
Overall Officials: Romulo A Fuentes Flores, PhD, Principal Investigator — University of Chile
Locations (1):
- Faculty of Medicine of University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No